CLINICAL TRIAL: NCT01375257
Title: Partial Oral Treatment of Endocarditis
Acronym: POET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kasper Iversen, Consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endocarditis-DK
Record Dates: First submitted 2011-06-13; First posted 2011-06-17 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Therapeutics; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guideline treatment with parenteral antibiotics (Active Comparator): Guideline treatment with parenteral antibiotics
  Interventions: Drug: Guideline treatment with parenteral antibiotics
- Oral treatment with antibiotics (Experimental): Oral treatment with antibiotics based on resistens pattern
  Interventions: Drug: Oral treatment with antibiotics for endocarditis

INTERVENTIONS:
Drug: Oral treatment with antibiotics for endocarditis
  Arms: Oral treatment with antibiotics
Drug: Guideline treatment with parenteral antibiotics
  Arms: Guideline treatment with parenteral antibiotics

SUMMARY:
Background Current management of infective endocarditis include admission and treatment with parenteral antibiotics for 4 weeks - 6 weeks. Resource demands and psychological issues of present management strategy make it highly relevant to seek for alternative more lenient alternatives. Experiences with oral treatment are only sporadically described, but observational data suggest that oral treatment could be a feasible option. The investigators have in 2010 treated 12 endocarditis patients with partial oral antibiotics with a 100% success rate.

Study design The POET study is a Danish multicenter, prospective, randomized, open label study. The primary aim is to show non-inferiority of partial oral treatment with antibiotics of endocarditis compared to full parenteral treatment. Stable patients (n=400) with streptococci, staphylococci or enterococci infecting the mitral valve or the aortic valve will be included. After a minimum of 10 days of parenteral treatment, patients will be randomized to oral therapy or parenteral therapy. Special recommendations for oral treatment have been developed based on expected minimal inhibitory concentrations and pharmacokinetic calculations. Patients will be followed for 6 months after completion of antibiotic therapy. The primary endpoint is a composition of all cause mortality, unplanned cardiac surgery, embolic events and relapse of positive blood cultures with the primary pathogen.

ELIGIBILITY:
Inclusion Criteria:

* Left-sided endocarditis based on the Duke criteria
* Infected with one of the following microorganisms:

  * Streptococci
  * Enterococcus faecalis
  * Staphylococcus aureus
  * Coagulase-negative staphylococci.
* ≥ 18 years
* At least 10 days of appropriate parenteral antibiotic treatment overall, and at least 1 week of appropriate parenteral treatment after valve surgery
* Afebrile (T < 38.0) > 2 days
* Decreasing infection parameters (CRP dropped to less than 25% of peak value or < 20 mg/l, and white blood cell count < 15 x 109/l) during antibiotic treatment
* No sign of abscess formation by echocardiography
* Transthoracic and transoesophageal echocardiography performed within 48 hours prior to randomization

Exclusion Criteria:

* Body mass index > 40
* Concomitant infection requiring intravenous antibiotic therapy
* Inability to give informed consent to participation
* Suspicion of reduced absorption of oral treatment due to abdominal disorder
* Reduced compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is a composite endpoint including all cause mortality, unplanned cardiac surgery, embolic events and relapse of positive blood cultures with the primary pathogen | Approximately 7 months. From randomisation until 6 months after end of study medication

SECONDARY OUTCOMES:
Quality of life | Approximately 7 months. From randomisation until 6 months after end of study medication
  QOL performed during the study and after completion of the study
Cost of treatment | Approximately 7 months. From randomisation until 6 months after end of study medication
Duration of antibiotic therapy | Approximately 7 months. From randomisation until 6 months after end of study medication
Complications related to intravenous catheter | 6 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- Denmark (8):
  - Aalborg Sygehus, Aalborg
  - Skejby Sygehus, Aarhus
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Copenhagen
  - Herlev Hoslpital, Copenhagen
  - Hillerød Hospital, Hillerød
  - Odense Sygehus, Odense
  - Roskilde Sygehus, Roskilde

REFERENCES:
- [Derived] Bundgaard JS, Iversen K, Pries-Heje M, Ihlemann N, Gill SU, Madsen T, Elming H, Povlsen JA, Bruun NE, Hofsten DE, Fuursted K, Christensen JJ, Schultz M, Rosenvinge F, Helweg-Larsen J, Kober L, Torp-Pedersen C, Fosbol EL, Tonder N, Moser C, Bundgaard H, Mogensen UM. Self-assessed health status and associated mortality in endocarditis: secondary findings from the POET trial. Qual Life Res. 2022 Sep;31(9):2655-2662. doi: 10.1007/s11136-022-03126-x. Epub 2022 Mar 29. PMID 35349038
- [Derived] Iversen K, Ihlemann N, Gill SU, Madsen T, Elming H, Jensen KT, Bruun NE, Hofsten DE, Fursted K, Christensen JJ, Schultz M, Klein CF, Fosboll EL, Rosenvinge F, Schonheyder HC, Kober L, Torp-Pedersen C, Helweg-Larsen J, Tonder N, Moser C, Bundgaard H. Partial Oral versus Intravenous Antibiotic Treatment of Endocarditis. N Engl J Med. 2019 Jan 31;380(5):415-424. doi: 10.1056/NEJMoa1808312. Epub 2018 Aug 28. PMID 30152252
- [Derived] Iversen K, Host N, Bruun NE, Elming H, Pump B, Christensen JJ, Gill S, Rosenvinge F, Wiggers H, Fuursted K, Holst-Hansen C, Korup E, Schonheyder HC, Hassager C, Hofsten D, Larsen JH, Moser C, Ihlemann N, Bundgaard H. Partial oral treatment of endocarditis. Am Heart J. 2013 Feb;165(2):116-22. doi: 10.1016/j.ahj.2012.11.006. Epub 2013 Jan 3. PMID 23351813